CLINICAL TRIAL: NCT01518829
Title: Role of Procalcitonin in Differantiation Between Bacerial Infection and Non Infectious Inflammation in Febrile Hepatocellular Carcinoma Patients After Locoregional Treatment
Brief Title: Procalcitonin in Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of Tropical medicine ,Faculty of Medicine,Ain Shams university, Ain Shams University
Other Study IDs: HCC and Procalcitonin
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinom; postablation syndrom; procalcitonin
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with hepatocellular carcinoma: Patients with hepatocellular carcinoma who will undergo locoregional therapy
- patients with chronic liver disease: patients with chronic liver disease, as a control group

SUMMARY:
the value of serum procalcitonin in differentiation between bacterial infection and non infectious inflammation in febrile HCC patients following locoeregional treatment for HCC.

ELIGIBILITY:
Inclusion Criteria:

1. - Hepatocellular carcinoma patients who will undergo TACE and/or radio-frequency.
2. - Fever more than 38C after 48 hours post intervention.

Exclusion Criteria:

1. HCC Patients who does not develop fever after intervention.
2. Proven infection elsewhere (e.g. UTI, chest infection..)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatients in tropical medicine department and hepatocellular carcinoma out patient clinic ain shams university
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Differantiate between post- embolization syndrom and sepsis following locoregional treatment for hepatocellular carcinoma | 6months

CONTACTS AND LOCATIONS:
Overall Officials: Hisham K Dabbous, professor, Principal Investigator — Tropical medicine department
Locations (1):
- Tropical medicine department and hepatocellular carcinoma clinic, Cairo, Egypt